CLINICAL TRIAL: NCT02127268
Title: Thymosin-α1 for Cancer-Related Fatigue in Cancer Patients Who Undergo Chemotherapy: A Randomized Controlled Trial
Brief Title: Thymosin-α1 in Cancer-Related Fatigue
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhigang Zhang (Other)
Responsible Party: Sponsor-Investigator, Zhigang Zhang, Doctor, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: T-CRF
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Cancer Related Fatigue; Quality of Life

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm T (Active Comparator): Will be treated with Thymosin-α1 1.6mg twice a week from day 1 of chemotherapy
  Interventions: Drug: Thymosin-α1
- Arm B (No Intervention): With best support according to NCCN Guideline

INTERVENTIONS:
Drug: Thymosin-α1 — with Thymosin-α1 1.6mg twice a week
  Arms: Arm T

SUMMARY:
Cancer-related fatigue (CRF) is a distressing, persistent, subjective sense of physical, emotional, and/or cognitive tiredness or exhaustion related to cancer or cancer treatment that is not proportion to recent activity and interferes with usual functioning. Compared with general fatigue, CRF have the characteristics of long duration and generally cannot alleviate by rest or sleep, serious impact on the patient's work, study, entertainment and family life, and thus greatly affect the recovery, self-care ability and life quality of patients. Many dates showed that 70%~100% of cancer patients experienced cancer-related fatigue.For cancer-related fatigue there is no good treatment and intervention, in recent years, many clinical trials are carried out; central nervous stimulant, such as methylphenidate; acupuncture, aerobic exercise. All those measures may have certain therapeutic effect for CRF, but don't have exact evidences from massive RCT to confirm.

Thymosin-α1 (T-α1), a synthetic 28-amino acid peptide with multiple biological activities primarily directed towards immune response enhancement, this drug is used for the treatment of HBV and hepatitis C virus (HCV) infections, and being developed for the treatment of non-small cell lung cancer (NSCLC), hepatocellular carcinoma, AIDS and malignant melanoma. T-α1 is able to potentiate the action of cytokines and also reduce the hematological toxicity of cytotoxic drug therapy, such as cyclophosphamide, 5-fluorouracil, dacarbazine.

In this studies, we want to demonstrated that the effectiveness of Thymosin-α1 for cancer-related fatigue in cancer patients who undergo chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 years and older.
2. The life expectancy at least 6 months.
3. With a definite pathological diagnosis of cancer, and undergo chemotherapy.
4. Patients who are willing to participate in the study.

Exclusion Criteria:

1. Thymosin-α1 allergy.
2. Using the spirit excitement or stimulant drugs.
3. With brain metastasis or primary malignant brain tumors.
4. With mental disorders, such as suffering from dementia, delirium, obsessive-compulsive disorder, schizophrenia, epilepsy.
5. Other specific causes of fatigue: such as anemia, thyroid function is low, insomnia, uncontrolled pain.
6. Serious HRS cardiopulmonary function disorder.
7. Women during pregnancy and lactation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in Cancer-Related Fatigue Scale | baseline and 4 weeks

SECONDARY OUTCOMES:
improvement in Quality of Life | baseline and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jian Huang, Doctor, Study Director — Zhejiang University
Locations (1):
- Cancer institute, Hangzhou, Zhejiang, China